CLINICAL TRIAL: NCT00883415
Title: A Study to Evaluate the Effect of the Treatment of Anemia on Myocardial Glucose Uptake (MGU) in Patients With Chronic Kidney Disease
Brief Title: Myocardial Glucose Uptake (MGU) in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Jeffrey Fink, Professor, Nephrology (primary); Epidemiology (secondary), University of Maryland, Baltimore
Other Study IDs: HP-00041025; Amgen ISS#20061907
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Cardiomyopathy; Chronic Kidney Disease; Anemia
Keywords: metabolism; myocardium; chronic kidney disease
MeSH Terms: conditions — Cardiomyopathies; Renal Insufficiency, Chronic; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Darbepoetin alfa — Subjects will undergo anemia management with darbepoetin after baseline assessment of MGU and will continue for six months with repeat assessment of MGU at completion of protocol
  Other Names: Aranesp

SUMMARY:
This study examines patients with chronic kidney disease-related anemia and measures changes in the metabolism of the heart using FDG/PET scanning, before and 6 months after their health-care provider has initiated anemia management therapy with the FDA-approved drug darbepoetin alfa (Aranesp), which is approved for chronic kidney disease-related anemia. The investigators hypothesize that the heart has abnormal metabolism with the anemia of chronic kidney disease but this improves after correction of this anemia with darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Participant must receive care at the VAMHCS (VA Hospital) in Baltimore
* Diagnosed with CKD stage 3 to 5 (eGFR of 60 ml/min/1.73m2) and not expected to initiate renal replacement therapy within 6 months
* Anemia related CKD.
* The last 2 serum hemoglobin (Hb) values less than 11.0 gm/dl but greater than 8.0 gm/dl
* Greater than 18 years of age
* Assessed to be clinically stable by the clinician

Exclusion Criteria:

* Need for hemodialysis, peritoneal dialysis, or transplantation at the time of enrollment or projected to start within 6 months after enrollment
* Low functional capacity including inability to walk a flight of stairs with a bag of groceries (NYHA Class III/IV Heart Failure)
* Prior erythropoietic agents within last 12 weeks
* TSAT < 15% and not receiving the recommended dose for iron deficiency
* Uncontrolled hypertension defined as greater than 180 mm Hg systolic or 110 mm Hg diastolic
* Potentially "brittle" diabetes with the propensity for symptomatic hypoglycemia after a 6 hour fast
* New diagnosis or ongoing therapy for Cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals being followed for their chronic kidney disease (CKD) at one of the Nephrology/Early Renal Insufficiency Clinics at the Baltimore, Maryland VA Medical Center and are being considered for erthropoietin therapy for anemia related to CKD.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Fink, MD MS, Principal Investigator — University of Maryland School of Medicine and Baltimore VA
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-post Intervention Evaluation: Changes in myocardial glucose uptake were evaluated in each participant before and after anemia treatment with darbepoetin alfa.
Period: Overall Study
Arm/Group | Pre-post Intervention Evaluation
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change to Myocardial Glucose Uptake as Measured by Fluoro-deoxy-D-glucose (FDG) Positron Emission Tomography (PET) Scan From Pre-treatment Compared to 6 Months After Anemia Therapy Initiation.
Description: Change in myocardial glucose uptake from baseline to 6 months expressed as change in micromol/min/100 g
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: micromol/min/100g
Arm/Group | Intervention
Number analyzed (Participants) | 18
micromol/min/100g | 4.49 [-6.75 to 15.73]

ADVERSE EVENTS:
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=20)
Gastric Carcinoma (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No